CLINICAL TRIAL: NCT05721443
Title: Cetuximab Plus Dalpicilib in the Second-line Treatment of Patients With HPV Negative, PD-1 Resistant Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma: an Open-label,Single Arm,Phase 2 Trial
Brief Title: Cetuximab Plus Dalpicilib in Patients With HPV Negative, PD-1 Resistant R/M HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2022-T252-1
Record Dates: First submitted 2022-11-09; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-10

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib+cetuximab (Experimental): The dosing regimen for cetuximab combined with dalpiciclib is: the starting dose of cetuximab is 400 mg/m2, titrated over 120 minutes, and the titration rate should be limited to 5 ml/min. A maintenance dose of 250 mg/m2, titrated over not less than 60 minutes, with pretreatment with H1 receptor blocker desensitization prior to dosing, administered once weekly.
  The recommended dose of dalpiciclib is 150 mg once daily for 21 days, followed by 7 days of discontinuation (3/1 dosing regimen) for a 28-day treatment cycle. Take the drug at approximately the same time each day. If the patient vomits or misses a dose, the dose should not be made up that day. The next dose should be taken as usual.
  Subjects will continue treatment with cetuximab in combination with dalpiciclib until termination criteria are met.
  Interventions: Drug: Dalpiciclib+cetuximab

INTERVENTIONS:
Drug: Dalpiciclib+cetuximab — The dosing regimen for cetuximab combined with dalpiciclib is: the starting dose of cetuximab is 400 mg/m2, titrated over 120 minutes, and the titration rate should be limited to 5 ml/min. A maintenance dose of 250 mg/m2, titrated over not less than 60 minutes, with pretreatment with H1 receptor blocker desensitization prior to dosing, administered once weekly.
  The recommended dose of dalpiciclib is 150 mg once daily for 21 days, followed by 7 days of discontinuation (3/1 dosing regimen) for a 28-day treatment cycle. Take the drug at approximately the same time each day. If the patient vomits or misses a dose, the dose should not be made up that day. The next dose should be taken as usual.
  Subjects will continue treatment with cetuximab in combination with dalpiciclib until termination criteria are met.

SUMMARY:
This study is the first clinical study in PD-1 resistant patients with head and neck squamous cell carcinoma with drugs targeting EGFR signaling pathway combined with CDK4/6 inhibitors, which explores the new combination therapies urgently needed in clinical practice and lays a foundation for subsequent studies, with important scientific research significance and clinical value.

DETAILED DESCRIPTION:
Head and neck cancer is the sixth most common cancer in the world, with more than 550,000 incidences and 300,000 deaths per year worldwide. more than 95% of head and neck cancers are squamous cell carcinomas, and head and neck squamous cell carcinoma (HNSCC) has a devastating and HNSCC affects the quality of life of patients by damaging and affecting their appearance and basic physical, sensory and speech functions. Due to the difficulty of early detection, more than 60% of head and neck squamous cell carcinoma patients are already at locally advanced stage when detected, and the prognosis of locally advanced head and neck carcinoma is poor, and even after receiving aggressive treatment, it is prone to local recurrence and distant metastasis after treatment.

About 25% of patients with squamous head and neck cancer are associated with human papillomavirus (HPV) infection, of which the most common subtype is HPV 16, accounting for more than 80% of all HPV-induced head and neck cancers. HPV infection suppresses the function of oncogenes TP53 and RB, and promotes immune escape and promote the development of head and neck cancer. In China, more than 70% of head and neck squamous carcinomas are not associated with HPV infection, and compared with HPV-associated HNSCC, HPV-negative HNSCC has a lower response rate to treatment and the overall prognosis of patients is worse.

Head and neck squamous cell carcinoma has a high rate of Treg cell as well as NK cell infiltration in the tumor microenvironment, forming an immunosuppressive tumor microenvironment and is a group of malignancies with high immunodeficiency. Studies have shown high levels of PD-L1 expression in tumor tissue in 46%-100% of HNSCC. Therefore, blockade of immune checkpoint inhibitors represented by PD-L1/PD-1 is a theoretically feasible therapeutic approach for the treatment of HNSCC. The results of previous clinical trials of immunotherapy in patients with recurrent or metastatic head and neck squamous carcinoma showed that anti-PD-1 antibodies led to durable remission and improved survival in patients with either first- or second-line therapy. The KEYNOTE-048 study confirmed that pembrolizumab in combination with chemotherapy prolonged overall survival in patients with recurrent or metastatic head and neck squamous carcinoma and in 2021 recommended by CSCO guidelines as a first-line expert recommendation for the first-line treatment of recurrent or metastatic head and neck squamous carcinoma (Level of Evidence 1A). However, patients with recurrent or metastatic head and neck squamous carcinoma after failure of first-line applied anti-PD-1 therapy enter second-line therapy The current guideline recommended second-line treatment regimens are cetuximab, afatinib or methotrexate, but the overall prognosis of patients is poor, the drug response rate is not high, the highest objective remission rate reported in the literature is only 13%, and the time to tumor progression is only 2.3 months, therefore, exploring new second-line treatment options for patients with recurrent or metastatic head and neck squamous carcinoma after failure of anti-PD-1 therapy is a pressing clinical need.

In addition, the results of previous clinical trials showed that HPV-negative HNSCC had poorer sensitivity and prognosis to immunotherapy than HPV-associated HNSCC. In KEYNOTE-012, patients with HPV-positive HNSCC had higher objective remission (32% vs 14%) and progression-free survival (4 months vs 2 months) with pablizumab, and similar results were confirmed by KEYNOTE-055. Furthermore, in a meta-analysis of 11 studies, HPV-positive HNSCC patients showed a 1.29-fold higher response rate to immunotherapy and a twofold higher overall survival (11.5 months vs. 6.3 months) than HPV-negative HNSCC patients.

There are a large number of ongoing clinical trials of combination targeted therapies and immunotherapies. The basic rationale supporting these combinations is that the two therapies combine different immunological and tumor biological mechanisms that enhance antitumor activity; in addition, some evidence suggests that targeted therapies can enhance certain aspects of the "cancer-immune cycle" (e.g., tumor antigenicity, T-cell initiation/transport/infiltration, etc.) to immunotherapy. In addition, it has been shown that targeted therapies can synergistically enhance certain aspects of the "cancer-immune cycle" (e.g., tumor antigenicity, T cell initiation/transport/infiltration, etc.) for immunotherapy. CDK4, one of the key cell cycle regulators, is involved in cell growth, proliferation, dormancy or apoptosis by binding to cell cycle protein D, which regulates the transition from G1 phase (pre-DNA synthesis) to S phase (DNA synthesis). In 2013, the US Food and Drug Administration (FDA) approved the CDK4 inhibitor Palbociclib as a breakthrough new drug for the treatment of advanced breast cancer, and the National Comprehensive Cancer Network (NCCN) guidelines recommend piperacillin in combination with an aromatase inhibitor as a first-line treatment option for HR+/HER2-advanced or metastatic breast cancer. Recent studies have found that CDK4 gene inhibition in combination with afatinib synergistically enhances the inhibition of the PI3k pathway in head and neck cancer cells, which in turn reduces tumor proliferation, providing a strong rationale for combination therapy.

P16 deletion is a hallmark event in HPV-negative HNSCC patients, and p16 inactivation would lead to CDK4/6 hyperactivation, making CDK4/6 theoretically a potential target for HPV-negative HNSCC. Some progress has been made with CDK4/6 inhibitors in HPV-negative head and neck squamous carcinoma. In a multicenter, multicohort phase II clinical trial, cohort 1 enrolled in first-line treatment of platinum-resistant HPV-negative patients with recurrent/metastatic HNSCC, and cohort 2 enrolled in first-line treatment of cetuximab-resistant HPV-negative cohort 3 enrolled patients with cetuximab-resistant HPV-positive recurrent/metastatic oropharyngeal cancer, and all three groups received Palbociclib in combination with cetuximab, showing objective remission rates of up to 39% in cohort 1 and 19% in cohort 2, but only 4% in cohort 3, indicating that CDK4/6 inhibitors in combination with cetuximab has a promising application in the treatment of HPV-negative HNSCC.

This clinical study involved dalpiciclib, which was developed by Jiangsu Hengrui Pharmaceutical Co. In December 2021, the State Drug Administration approved the drug in combination with fulvestrant for patients with recurrent or metastatic breast cancer with hormone receptor-positive, human epidermal growth factor receptor 2-negative disease progression after previous endocrine therapy through a priority review and approval process. Patients. Preclinical studies have shown that dalpiciclib has comparable in vivo efficacy and safety compared to its foreign counterparts.

This study is also the first clinical study of a drug targeting CDK4/6 in combination with cetuximab for the treatment of HPV-negative head and neck squamous carcinoma after progression of PD-1 therapy in China, which is of great scientific significance and clinical value in exploring new combination therapies for HPV-negative patients, a population with poor clinical outcome, and laying the foundation for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, both sexes.
* Patients with histologically confirmed post-surgical recurrent/metastatic or locally advanced inoperable surgically resectable squamous cell carcinoma of the head and neck with measurable lesions (spiral CT scan ≥ 10 mm, meeting RECIST 1.1 criteria).
* Have received at least 1 cycle of prior PD-1 immunotherapy with imaging confirmation of progression or clinician determination of no continued benefit from treatment; provided that this is completed at least 4 weeks prior to the first dose of study drug and all associated toxic events have returned to normal or grade I or less as defined by CTCAE 4.03 classification.
* HPV viral testing determined to be negative, using the IHC method.
* Availability of tumor tissue (paraffin specimens less than 2 years old or fresh tumor tissue) for detection of PD-L1 and CDK4-related genes.
* ECOG score of 0 or 1.
* Expected survival of ≥ 12 weeks.
* Normal major organ function within 2 weeks prior to treatment, i.e., meeting the following criteria：Bone marrow function: hemoglobin ≥ 100 g/L without transfusion or colony-stimulating factor support therapy, white blood cell count ≥ 4.0*10^9/L or neutrophil count ≥ 2.0*10^9/L, and platelet count ≥ 100*10^9/L; Liver: serum total bilirubin level ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal; Renal: blood creatinine level below 1.5 times the upper limit of normal or creatinine clearance ≥ 60 ml/min and urea nitrogen ≤ 200 mg/L; Urine protein <+, or if urine protein + then total 24-hour protein must be <500mg; Blood glucose: within normal range and/or with diabetes in treatment but under stable glycemic control; Pulmonary function: baseline FEV1 of at least 2L; if baseline FEV1 <2L then FEV1 >800ml expected post-surgery as assessed by a surgical specialist; Cardiac function: no myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmias; no cardiac insufficiency.

Exclusion Criteria:

* Patients previously treated with cetuximab or other anti-EGFR monoclonal antibodies or small molecule tyrosine kinase inhibitors.
* Patients who are currently receiving antineoplastic therapy.
* Patients who have participated or are participating in a clinical trial of another drug/therapy within 4 weeks prior to the first dose of the study drug.
* Patients who have received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc., within 1 week prior to the first dose of the study drug.
* Positive HIV antibody or syphilis spirochete antibody test results.
* Patients with active hepatitis B or C: If positive for HBsAg or HBcAb, additional HBV DNA testing (results above the upper limit of the normal range). If HCV antibody test result is positive, add HCV RNA test (result above the upper limit of the normal range).
* Known hypersensitivity to recombinant humanized EGFR monoclonal antibody drugs and their components.
* Massive pleural or ascites fluid with clinical symptoms and requiring symptomatic management.
* Active lung disease (interstitial pneumonia, pneumonia, obstructive lung disease, asthma) or a history of active tuberculosis.
* Has any uncontrollable clinical problem, including but not limited to: Persistent or active (severe) infection; Poorly controlled diabetes mellitus; Cardiac disease (Class III/IV congestive heart failure or heart block as defined by the New York Heart Association); Deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism within 6 months prior to first dose.
* Previous stem cell transplantation or organ transplantation.
* Those with a history of psychotropic substance abuse and unable to abstain or a history of psychiatric disorders.
* Other serious, acute or chronic medical conditions or abnormalities in laboratory tests that, in the judgment of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Patients who, in the judgment of the investigator, have poor compliance or other conditions that make them unsuitable for participation in this trial.
* Patients with a history of other malignancies within five years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 24 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR:
  disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
overall survival | 24 months
  OS was defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Progression Free Survival Per RECIST 1.1 | 24 months
  PFS was defined as the time from enrollment to the first documented PD per RECIST 1.1, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD
Number of Participants Experiencing an Adverse Event (AE). | 24 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.
Quality of life#EORTC QLQ-C30 scale# | 24 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No